CLINICAL TRIAL: NCT00638872
Title: Diabetic Foot Ulcers and Use of PDRN (Polydeoxyribonucleotide -Placentex Mastelli) as a Treatment for Wound Healing.
Brief Title: Polydeoxyribonucleotide -Placentex Mastelli(Pdrn) for the Treatment of Diabetic Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Francesco Squadrito, Full Professor of Pharmacology, University of Messina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLA/01/06
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Diabetic Ulcer; Foot Ulcer Unhealed
Keywords: diabetes; foot ulcer; polydeoxyribonucleotide
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer | interventions — Polydeoxyribonucleotides; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): PDRN
  Interventions: Drug: Polydeoxyribonucleotide
- placebo (Placebo Comparator): placebo
  Interventions: Other: 0.9% NaCl

INTERVENTIONS:
Drug: Polydeoxyribonucleotide — 3 times a week perilesional or intramuscular injections
  Arms: 1
Other: 0.9% NaCl — same as PDRN
  Arms: placebo

SUMMARY:
The main objective of the study is to evaluate the efficacy of the polydeoxyribonucleotide in improving the healing of diabetic foot ulcers.

DETAILED DESCRIPTION:
This trial will involve diabetic patients with foot ulcers who meet the inclusion/exclusion criteria. At least 200 patients aged 45-80yrs will be enrolled in the study and randomly allocated to receive the active drug or the placebo in indistinguishable formulations. After 2 months closure rate of the ulcer will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 45-80yrs
* Minimum schooling 5yrs
* Type I or II diabetes since at least 5yrs with a stable metabolic control
* Foot ulcer since minimum 2 weeks
* Ulcer >1cm and <16cm at day 0
* Ulcer grade 1 or 2 wagner scale
* Wound free of necrotic debris
* TcPO2 >29mmHg
* Not pregnant or lactant

Exclusion Criteria:

* Non-consenting patient
* History of alcohol or drug abuse
* Gangrene on any part of the affected foot
* Ongoing untreated infections
* Ulcer over a charcot deformity
* Use of a systemic cicatrizant drug in the past 10 days
* Malnutrition
* Neurological or psychiatric pathologies
* Liver or kidney insufficiency
* Corticosteroid or immunosuppressive or cytotoxic therapy
* Other severe pathologies
* Proven hypersensitivity to the drug or to any related component

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2007-10; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
reduction of ulcer rate | 3 months

SECONDARY OUTCOMES:
safety and tolerability of the compound | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Cattarini, Study Director — Mastelli srl, via Bussana Vecchia, Sanremo, Italy
Locations (1):
- University of Messina, Messina, Italy